CLINICAL TRIAL: NCT02856295
Title: anti10a Levels in Women Treated With LMWH in the Postpartum Period for Preventing Vein Thrombosis Events: A Comparison of Two Doses
Brief Title: anti10a Levels in Women Treated With LMWH in the Postpartum Period
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Zohar Nachum, MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EMC59-12
Record Dates: First submitted 2016-07-13; First posted 2016-08-04 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Venous Thromboembolism
Keywords: postpartum venous thromboembolism; prophylactic dose of low molecular weight heparin; anti 10a
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clexane according to weight group (Active Comparator): clexane dose adjusted for woman's weight according to: weight < 90 kg - 40mg, 91-130kg - 60 mg, 131-170kg - 80mg, >170kg-100mg.
  Interventions: Drug: clexane (LMWH)
- clexane mg per kg (Active Comparator): clexane dose of 1mg/kg up to 120 mg
  Interventions: Drug: clexane (LMWH)

INTERVENTIONS:
Drug: clexane (LMWH) — to compare tow doses of clexane for preventing VTE in postpartum women

SUMMARY:
The aim of this study is to compare between anti-10a levels in postpartum women receiving different prophylactic doses of LMWH: one group with LMWH doses adjusted by the women's weight and the second group receiving 1mg/kg to a maximum dose of 120 mg

DETAILED DESCRIPTION:
pregnancy and postpartum period are associated with increased risk of thromboembolism. this risk is further increased in women with thrombophilia.

This risk is higher in the postpartum period compared with pregnancy period, especially the risk for pulmonary embolism (PE). The American College Of Obstetrics and Gynecologists, The American college of chest physicians and The Royal College of obstetricians and gynecologists recommend using low molecular weight heparin during the postpartum period in women with thrombophilia and women with risk factor for developing thromboembolism. there is no specific guidelines regarding the best protocol based on the level of anti-10 a.

This study will compare between two protocols based on anti-10a levels.

ELIGIBILITY:
Inclusion Criteria:

* postpartum women supposed to receive LMWH according to obstetric indications

Exclusion Criteria:

* known allergy to clexane
* active bleeding postpartum
* thrombocytopenia < 75000
* recent cerebrovascular accident / transient ischemic attack (<4 weeks)
* glomerular filtration rate) < 30 ml/min)
* active liver disease
* malignant hypertension (systolic > 200 mmHg, diastolic> 120 mmHg)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
clexane dosing method in order to achieve anti 10a level >0.2 | 4 hour after the women receive the drug

SECONDARY OUTCOMES:
incidence of anti 10a level of >0.6 | 4 hour after the women receive the drug
incidence of vein thromboembolism | during the six weeks after delivery
incidence of bleeding events | during the six weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Nachum, M.D, Study Director — Emek Medical Center
Locations (1):
- Emek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bremme KA. Haemostatic changes in pregnancy. Best Pract Res Clin Haematol. 2003 Jun;16(2):153-68. doi: 10.1016/s1521-6926(03)00021-5. PMID 12763484
- [Result] Hellgren M. Hemostasis during normal pregnancy and puerperium. Semin Thromb Hemost. 2003 Apr;29(2):125-30. doi: 10.1055/s-2003-38897. PMID 12709915
- [Result] Practice bulletin no. 124: inherited thrombophilias in pregnancy. Obstet Gynecol. 2011 Sep;118(3):730-740. doi: 10.1097/AOG.0b013e3182310c6f. PMID 21860314
- [Result] Scifres CM, Macones GA. The utility of thrombophilia testing in pregnant women with thrombosis: fact or fiction? Am J Obstet Gynecol. 2008 Oct;199(4):344.e1-7. doi: 10.1016/j.ajog.2008.04.051. Epub 2008 Jun 24. PMID 18572147
- [Result] Gherman RB, Goodwin TM, Leung B, Byrne JD, Hethumumi R, Montoro M. Incidence, clinical characteristics, and timing of objectively diagnosed venous thromboembolism during pregnancy. Obstet Gynecol. 1999 Nov;94(5 Pt 1):730-4. doi: 10.1016/s0029-7844(99)00426-3. PMID 10546719
- [Result] Chang J, Elam-Evans LD, Berg CJ, Herndon J, Flowers L, Seed KA, Syverson CJ. Pregnancy-related mortality surveillance--United States, 1991--1999. MMWR Surveill Summ. 2003 Feb 21;52(2):1-8. PMID 12825542
- [Result] Heit JA, Kobbervig CE, James AH, Petterson TM, Bailey KR, Melton LJ 3rd. Trends in the incidence of venous thromboembolism during pregnancy or postpartum: a 30-year population-based study. Ann Intern Med. 2005 Nov 15;143(10):697-706. doi: 10.7326/0003-4819-143-10-200511150-00006. PMID 16287790
- [Result] Pomp ER, Lenselink AM, Rosendaal FR, Doggen CJ. Pregnancy, the postpartum period and prothrombotic defects: risk of venous thrombosis in the MEGA study. J Thromb Haemost. 2008 Apr;6(4):632-7. doi: 10.1111/j.1538-7836.2008.02921.x. Epub 2008 Jan 31. PMID 18248600
- [Result] McColl MD, Walker ID, Greer IA. The role of inherited thrombophilia in venous thromboembolism associated with pregnancy. Br J Obstet Gynaecol. 1999 Aug;106(8):756-66. doi: 10.1111/j.1471-0528.1999.tb08395.x. PMID 10453824
- [Result] Bates SM, Greer IA, Middeldorp S, Veenstra DL, Prabulos AM, Vandvik PO. VTE, thrombophilia, antithrombotic therapy, and pregnancy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e691S-e736S. doi: 10.1378/chest.11-2300. PMID 22315276
- [Result] American College of Obstetricians and Gynecologists. ACOG Committee Opinion: safety of Lovenox in pregnancy. Obstet Gynecol. 2002 Oct;100(4):845-6. PMID 12387283
- [Result] Bain E, Wilson A, Tooher R, Gates S, Davis LJ, Middleton P. Prophylaxis for venous thromboembolic disease in pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2014 Feb 11;(2):CD001689. doi: 10.1002/14651858.CD001689.pub3. PMID 24519568
- [Result] Bates SM, Greer IA, Hirsh J, Ginsberg JS. Use of antithrombotic agents during pregnancy: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):627S-644S. doi: 10.1378/chest.126.3_suppl.627S. PMID 15383488
- [Result] Shapiro NL, Kominiarek MA, Nutescu EA, Chevalier AB, Hibbard JU. Dosing and monitoring of low-molecular-weight heparin in high-risk pregnancy: single-center experience. Pharmacotherapy. 2011 Jul;31(7):678-85. doi: 10.1592/phco.31.7.678. PMID 21923455
- [Result] Fox NS, Laughon SK, Bender SD, Saltzman DH, Rebarber A. Anti-factor Xa plasma levels in pregnant women receiving low molecular weight heparin thromboprophylaxis. Obstet Gynecol. 2008 Oct;112(4):884-9. doi: 10.1097/AOG.0b013e31818638dc. Erratum In: Obstet Gynecol. 2009 Mar;113(3):742. PMID 18827132
- [Derived] Haj R, Massalha M, Eitam H, Kassabri R, Yefet E, Nachum Z. Comparison of postpartum anti-Xa levels following enoxaparin administration to prevent venous thromboembolism using 2 weight-based protocols: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Aug;5(8):100988. doi: 10.1016/j.ajogmf.2023.100988. Epub 2023 May 6. PMID 37156466